CLINICAL TRIAL: NCT06814054
Title: Carotid Artery Corrected Flow Time and Inferior Vena Cava Collapsibility Index for Prediction of Hypotension After Induction of General Anesthesia in Geriatric Patients Undergoing Elective Surgery
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Other Study IDs: Hypotension in geriatrics
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Geriatrics; Hypotension on Induction; General Anesthetic Drug Adverse Reaction; Elective Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GA induced hypotension in geriatrics: Postinduction hypotension will be defined as either
  * A 30% drop in SBP or 20% drop in MAP from baseline, or an absolute SBP of less than 90 mm Hg and MAP of less than 65 mm Hg within three minutes of general anaesthesia induction, every minute until 15 min after endotracheal intubation and before the start of any surgical manipulations.
  * Since endotracheal intubation and direct laryngoscopy can generate sympathetic activation, which will change blood pressure, we decided to start haemodynamic monitoring three minutes post endotracheal intubation.
  * If the MAP was less than 65 mmHg, a 250 ml crystalloid bolus will be administered and repeated as necessary.
  * If hypotension persist after IV fluid bolus, ephedrine will be given by three milligrams.
  At the end of surgery.
  Interventions: Diagnostic Test: Carotid Artery Corrected Flow Time measurement; Diagnostic Test: Inferior vena cava collapsibility index

INTERVENTIONS:
Diagnostic Test: Carotid Artery Corrected Flow Time measurement — * The cFT is defined as the time between the onset of systolic flow until closure of the aortic valve corrected for the HR and has been found to correlate with the intravascular volume.
  * carotid ultrasound imaging will be performed 10 minutes before induction of general anesthesia in the preoperative holding area.
  * Ultrasound measurements will be performed under a vascular setting with a 6.0 to 13.0MHz linear array transducer
  * The right common carotid artery cFT will be measured in supine position with their heads tilted 30° to the left
  * After that, a pulse wave Doppler will be chosen, and the sampling frame will be positioned at an angle of less than 60° in the region of the carotid artery with the best color flow to acquire the blood flow spectrum.
Diagnostic Test: Inferior vena cava collapsibility index — * The IVC will be examined while the patient has been spontaneously, quietly breathing and lying in the supine position for at least 5 min before assessment.
  * A two-dimensional image of the IVC as it entered the right atrium will be obtained through the paramedian long-axis view via a subcostal approach using a curvilinear phased array probe (2-5 MHz)
  * Then, using M-mode imaging produced at a medium sweep speed, changes in IVC diameter with breathing will be evaluated 2 to 3 cm distal to the right atrium.
  * During the same respiratory cycle, measurements will be made of the IVC's greatest expiratory diameter (dIVC expiration) and lowest inspiratory diameter (dIVC inspiration). The formula IVCCI = (dIVC expiration - dIVC inspiration) × 100/dIVC expiration will be used to determine IVCCI as a percentage. (12)
  * IVCCI will be assessed by the same trained anesthesiologist who was blinded to postin duction hemodynamic measurements.

SUMMARY:
In this observational study, we will assess cFT by Carotid ultrasound and IVC collapsibility index for prediction of hypotension after induction of general anesthesia in geriatric patients undergoing elective surgery.

DETAILED DESCRIPTION:
Following the onset of general anesthesia, hypotension is frequently observed, and intraoperative hypotension is linked to end organ damage following surgery, including cardiac ischemia and severe renal injury. postoperative end-organ damage depends on the duration and magnitude.

The incidence of hypotension after induction of general anesthesia varies and is influenced by the induction agent, patient characteristics, and the definition of hypotension.

Hypotension was defined by a 30% reduction in the SBP or 20% reduction in the MAP from baseline or an absolute SBP of less than 90 mm Hg and MAP of less than 65 mm Hg within 3 minutes after induction of general anesthesia.

Elderly people are more likely to experience hemodynamic fluctuation and hypotension due to the high prevalence of left ventricular diastolic failure, lower vascular reactivity and higher sensitivity to anesthetics. More significantly, older patients can't tolerate hypotension for a long time.

A variety of hemodynamic monitoring techniques have been used to predict post- anesthetic hypotension. Non-invasive cardiometry, ultrasound evaluation of fluid status, and pulse oximetry variables, such as the perfusion index and pulse variability index, were utilized.

Zhang and Critchley demonstrated that preoperative hypovolemia predicted postinduction hypotension as determined by the inferior vena cava (IVC) diameter and IVC collapsibility index.

In many clinical situations, volume-responsive patients have been identified using Doppler-derived metrics such as the peak blood flow peak velocity variation (ðVpeak) and the common carotid artery corrected flow time (cFT).

The carotid artery Doppler measures provide several benefits, including being noninvasive and being technically simple to obtain due to the carotid artery's superficial nature. Since the common carotid artery cFT is unaffected by respiratory attempts, it can also be used to assess a patient's volume responsiveness when they are breathing on their own.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists Physical Status I to Ⅱ
* receiving general anesthesia for elective surgery
* fasted for at least 6 to 8 hours were recruited in this study

Exclusion Criteria:

* • patients who refused to participate in the study

  * American Society of Anaesthesiologists Physical Status Ⅲ or Ⅳ
  * Patients with a history of peripheral arterial diseases or atherosclerosis
  * Patients with body mass index of greater than 30 kg/m2
  * Patients with arrhythmia or cardiomyopathy
  * Chronic obstructive pulmonary disease (COPD)
  * baseline systolic arterial pressure (SAP) ≥ 180 mmHg or < 90mmHg
  * Any episode of desaturation or difficult intubation during general anasethia induction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: geriatric patients (65 years and above) (10) of either sex and ASA PS I to Ⅱ receiving general anesthesia for elective surgery, who fasted for at least 6 to 8 hours were recruited in this study
Sampling Method: Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
the diagnostic efficacy of cFT by Carotid ultrasound and IVC collapsibility index in prediction of hypotension after induction of general anesthesia in geriatric patients | immediate preoperative peroid before the induction of general anesthesia
  the diagnostic efficacy of cFT by Carotid ultrasound and IVC collapsibility index in prediction of hypotension after induction of general anesthesia in geriatric patients undergoing elective surgery.

CONTACTS AND LOCATIONS:
Overall Officials: tarek Mostafa, Principal Investigator — tanta university, faculty of medicine
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No